CLINICAL TRIAL: NCT01535469
Title: Operational Research for Cryptococcal Antigen Screening to Improve ART Survival
Brief Title: Operational Research for Cryptococcal Antigen Screening
Acronym: ORCAS
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Infectious Diseases Institute, Uganda (Other); Makerere University (Other); Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: HS1254; U01GH000517 (NIH)
Record Dates: First submitted 2012-02-10; First posted 2012-02-17 (Estimated); Last update posted 2020-06-04 (Actual); Status verified 2020-06

CONDITIONS: Cryptococcal Meningitis; Cryptococcus Neoformans; Cryptococcosis
Keywords: cryptococcal meningitis; hiv; aids; implementation science; stepped wedge design; retention-in-care
MeSH Terms: conditions — Meningitis, Cryptococcal; Cryptococcosis; Acquired Immunodeficiency Syndrome | interventions — Fluconazole

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- CrAg Screening and Fluconazole (Experimental): Cryptococcal Antigen (CrAg) Screening with preemptive antifungal treatment per World Health Organization (WHO) guidelines. Randomized Stepped Wedge design of phased implementation.
  Interventions: Drug: Fluconazole

INTERVENTIONS:
Drug: Fluconazole — Fluconazole 800mg orally daily for 2 weeks, then 400mg daily for 8 weeks
  Other Names: Diflucan

SUMMARY:
This will be a stepped wedge randomized trial design to evaluate the implementation of cryptococcal antigen (CRAG) screening and preemptive anti-fungal therapy of HIV-infected persons entering antiretroviral therapy (ART) outpatient treatment in Uganda. Those who are ART eligible with a CD4≤100 cells/mcL will have a serum/plasma CRAG performed by lateral flow assay. Those who are CRAG-positive and asymptomatic will be treated with high dose fluconazole. After 6 months survival with retention-in-care will be compared between those who are CRAG+ and CRAG negative

ELIGIBILITY:
Inclusion Criteria:

* HIV-1 infection
* CD4≤100 cells/mcL
* Cryptococcal antigen (CRAG) positive
* age >14 years

Exclusion Criteria:

* Suspected Cryptococcal meningitis
* Prior known history of cryptococcal meningitis
* currently receiving HIV antiretroviral therapy
* Allergy to any azole antifungal medication
* Persons with known serious hepatic co-morbidities, transaminitis, or clinical jaundice who should not receive fluconazole in the opinion of the study investigator.
* Current known pregnancy

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 3049 (Actual)
Dates: Start 2012-07-01 (Actual); Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Retention in care | 6-month
  1. before/after CRAG screening implementation (All persons)
  2. CRAG positive persons treated with high-dose fluconazole as compared to 6-month survival of CRAG negative persons who are eligible for antiretroviral therapy.

SECONDARY OUTCOMES:
Cryptococcal meningitis-free survival time | 6-month
  Cryptococcal meningitis-free survival time in those who are asymptomatic CRAG positive and treated with fluconazole compared to CRAG-negative persons with CD4<100 cells/mcL
Survival Time | 6-month
  Survival time among CRAG+ vs. CRAG negative persons with CD4<100 cells/mcL.
Uptake of CRAG screening and preemptive treatment | baseline
Time from CRAG+ test to receipt of fluconazole therapy | Days from CD4 testing
All-cause discontinuation of fluconazole | 6-month
  Number of participants with early discontinuation of fluconazole for any reason (e.g. non-compliance, adverse event)
Percentage of participants with symptomatic cryptococcal meningitis | baseline
Risk factors for symptomatic cryptococcal meningitis | baseline

CONTACTS AND LOCATIONS:
Overall Officials: David B Meya, MMed, Principal Investigator — Makerere University; Radha Rajasingham, MD, Study Director — Infectious Disease Institute
Locations (2):
- Uganda (2):
  - Infectious Disease Institute, Makerere University, Kampala
  - Kampala Capital Council Authority Clinics, Kampala

IPD SHARING:
Plan to Share IPD: Yes
After publication, data to be shared upon request to the Infectious Disease Institute Research Department as per the institutional data sharing policy.
Supporting Information: Study Protocol
Time Frame: Upon request
Access Criteria: Upon request

REFERENCES:
- [Background] Rajasingham R, Meya DB, Boulware DR. Integrating cryptococcal antigen screening and pre-emptive treatment into routine HIV care. J Acquir Immune Defic Syndr. 2012 Apr 15;59(5):e85-91. doi: 10.1097/QAI.0b013e31824c837e. PMID 22410867
- [Background] Meya DB, Manabe YC, Castelnuovo B, Cook BA, Elbireer AM, Kambugu A, Kamya MR, Bohjanen PR, Boulware DR. Cost-effectiveness of serum cryptococcal antigen screening to prevent deaths among HIV-infected persons with a CD4+ cell count < or = 100 cells/microL who start HIV therapy in resource-limited settings. Clin Infect Dis. 2010 Aug 15;51(4):448-55. doi: 10.1086/655143. PMID 20597693
- [Result] Meya DB, Kiragga AN, Nalintya E, Morawski BM, Rajasingham R, Park BJ, Mubiru A, Kaplan JE, Manabe YC, Boulware DR. Reflexive Laboratory-Based Cryptococcal Antigen Screening and Preemptive Fluconazole Therapy for Cryptococcal Antigenemia in HIV-Infected Individuals With CD4 <100 Cells/microL: A Stepped-Wedge, Cluster-Randomized Trial. J Acquir Immune Defic Syndr. 2019 Feb 1;80(2):182-189. doi: 10.1097/QAI.0000000000001894. PMID 30399034
- See also: Infectious Disease Institute — http://www.idi-makerere.com